CLINICAL TRIAL: NCT06748313
Title: Grand Challenges Fermented Food - Achars (fermented Pickles) in Pakistan
Brief Title: Fermented Food - Achars (fermented Pickles) in Pakistan
Acronym: FF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Dr Syed Asad Ali, Professor, Aga Khan University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 51952
Record Dates: First submitted 2024-12-05; First posted 2024-12-27 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Maternal Health; Gut Health
Keywords: women of reproductive age; pregnant women; malnourished children; pakistan; microbiome; Fermented Foods; Fermented Achar; Fermented Pickle; Fermented Pickle - Achar

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- G1= Mango Pickle (Water-Based) (Experimental): This group will use 50 grams of Mango Pickle (Water-Based) daily as an intervention.
  Interventions: Other: Mango Pickle (Water-Based)
- G2= Mango Pickle (Oil Based) (Experimental): This group will use 50 grams of Mango Pickle (oil-based) daily as an intervention.
  Interventions: Other: Mango Pickle (Oil Based)
- G3= Carrot Pickle (Water-Based) (Experimental): This group will use 50 grams of Carrot Pickle (Water-Based) daily as an intervention.
  Interventions: Other: Carrot Pickle (Water-Based)
- G4= Radish Pickle (Water-Based) (Experimental): This group will use 50 grams of Radish Pickle (Water-Based) daily as an intervention.
  Interventions: Other: Radish Pickle (Water-Based)
- G5= Onion Pickle (Water-Based) (Experimental): This group will use 50 grams of Onion Pickle (Water-Based) daily as an intervention.
  Interventions: Other: Onion Pickle (Water-Based)
- G6= Lemon & Chili Pickle (Water-Based) (Experimental): This group will use 50 grams of Lemon & Chili Pickle (Water-Based) daily as an intervention.
  Interventions: Other: Lemon & Chili Pickle (Water-Based)
- Control (non-fermented vegetables or fruits) (No Intervention): This group will serve as "Control" (non-fermented vegetables or fruits).

INTERVENTIONS:
Other: Mango Pickle (Water-Based) — The ingredients used in Mango Pickle (Water-based) are Raw mangoes, Carrots, Lemon, Green chili, Gum Berry (Lasora), Grewia asiatica (Phalsa), Sea salt, Fenugreek seeds whole, Fenugreek mashed, Fennel seeds, Chili flakes, Coriander seeds, Turmeric powder, Cumin, Black seeds, Bay leaves, Mashed garlic, Mustard oil, Vinegar, and Water. The pickle's fermentation process will be completed in 6-7 days, and it will be ready to use.
  Other Names: Mango Achar
  Arms: G1= Mango Pickle (Water-Based)
Other: Mango Pickle (Oil Based) — The ingredients used in Mango Pickle (Oil-based) are Raw mangoes, Carrots, Lemon, Green chili, Gum Berry (Lasora), Grewia asiatica (Phalsa), Sea salt, Fenugreek seeds whole, Fenugreek mashed, Fennel seeds, Chili flakes, Coriander seeds, Turmeric powder, Cumin, Black seeds, Bay leaves, Vinegar, Mashed garlic, and Mustard oil. The pickle's fermentation process will be completed in 6-7 days, and it will be ready to use.
  Other Names: Mango Achar
  Arms: G2= Mango Pickle (Oil Based)
Other: Carrot Pickle (Water-Based) — The ingredients used in Carrot Pickle (Water-Based) are Carrots, Spring garlic, Turmeric, water, mashed mustard seeds, chili powder, salt, and Mustard oil. The pickle's fermentation process will be completed in 2-3 days, and it will be ready to use.
  Other Names: Carrot Achar
  Arms: G3= Carrot Pickle (Water-Based)
Other: Radish Pickle (Water-Based) — The ingredients used in Radish Pickle (Water-Based) are Radish, Spring garlic, Turmeric, water, mashed mustard seeds, chili powder, salt, and Mustard oil. The pickle's fermentation process will be completed in 2-3 days, and it will be ready to use.
  Other Names: Radish Achar
  Arms: G4= Radish Pickle (Water-Based)
Other: Onion Pickle (Water-Based) — The ingredients used in Onion Pickle (Water-Based) are Onion, Vinegar, Turmeric, water, mashed mustard seeds, chili powder, salt, and Mustard oil. The pickle's fermentation process will be completed in 3-4 days, and it will be ready to use.
  Other Names: Onion Achar
  Arms: G5= Onion Pickle (Water-Based)
Other: Lemon & Chili Pickle (Water-Based) — The ingredients used in Lemon & Chili Pickle (Water-Based) are Lemon, Green Chili, Turmeric, Vinegar, water, and salt. The pickle's fermentation process will be completed in 2-3 days, and it will be ready to use.
  Other Names: Lemon Achar
  Arms: G6= Lemon & Chili Pickle (Water-Based)

SUMMARY:
The highest burden of malnutrition in the world is in South Asia and Africa. Over the last ten years, our work on Environmental Enteric Dysfunction in Matiari, a poor rural district in the Sind province of Pakistan, shows that the most critical driver of childhood stunting is anthropometry at birth. Birth anthropometry is primarily influenced by maternal health and nutrition. Fermented foods are an indigenous yet underutilized resource that could improve gut health, reduce inflammation, and promote a healthy microbiome in women. The most common plant-based fermented food used in rural Sind is the achar, a local variety of fermented pickles made from many different vegetables and fruits. Achar has been used over centuries in this area. Traditional folklore dictates that achar is good for pregnancy. Craving for achar is a sign of early pregnancy in this culture. Achars are considered antiemetics and are believed to help relieve gastric issues in early pregnancy.

The medical benefits of pickles/achars are fairly well recognized. Major microbes involved in the fermentation of Achar are LAB (Lactic Acid Bacteria), bacillus, and micrococcus species, which are directly or indirectly responsible for multiple health benefits. However, a clinical trial has not been conducted to determine the impact of regular use of achar on the health of women of childbearing age in a real-life setting.

The investigator hypothesizes that traditional, fermented achar use reduces gut and systemic inflammation and drives a healthy microbiome in women of reproductive age in Matiari, rural Sindh, Pakistan. If our trial confirms this hypothesis, then at-scale use of the best achars can be advocated in this community as an Indigenous and culturally appropriate intervention.

DETAILED DESCRIPTION:
The investigator recruited 210 women of reproductive age (18-45 years), including pregnant women. These women were divided into seven groups. Six groups were randomly assigned as "Test," and one group served as "Control" (non-fermented vegetables or fruits). Different formulations of achar were assigned to each of the groups.

G1= Mango Pickle (Water-Based) G2= Mango Pickle (Oil Based) G3= Carrot Pickle (Water-Based) G4= Radish Pickle (Water-Based) G5= Onion Pickle (Water-Based) G6= Lemon & Chili Pickle (Water-Based)

Women were recruited from the community through a demographic surveillance system established in Matiari, Pakistan. The study staff approached and introduced the potential participants to this study. If Participants agree, After informed consent, a short questionnaire was filled out, including information about socio-demographics, household food insecurity index, history of illness, and anthropometric measurements. 10ml blood samples were collected at baseline and at 8 weeks. 5ml blood sample was used for CBC and cytokine measurement while 5ml blood was required to collect PBMCs which was used for Transcriptomics analyses as complete immune-profiling is necessary to study the microbiome-host interaction and its impact on immune cells. Fecal samples were collected longitudinally for biomarkers assessment and fecal microbiome at baseline, at 8 weeks, and then at 12 weeks. A 24-hour food recall form was filled out at enrollment and at 8 weeks. We delivered pickles to the intervention group. The investigator did not offer anything for the control group. However, control participants were requested to eat non-fermented food and avoid fermented foods. The investigator collected information about compliance with treatment (Test group) after every 14 days. Common food items consumed in the last 7 days were collected through the food frequency form at each follow-up. Participants in intervention groups were given pickles in 50 gms of pre-weighted cups/jars for daily consumption, and partially eaten pickle cups were weighed again at each follow-up to measure compliance and standardization of pickle intake. All jars will be bar-coded. The study team will ensure the refilling of pickles at the household level.

ELIGIBILITY:
Inclusion Criteria:

• Women of reproductive age group (18-49 years) residing in the study area and should provide informed consent for study participation.

Exclusion Criteria:

* Antibiotics or probiotics or laxatives use in the past two weeks.
* Current diarrheal illness.
* Regular (>= two times a week) use of achars before enrollment.
* Any Gastrointestinal illness such as chronic constipation, Irritable bowel syndrome, Gastroesophageal Reflux Disease (GERD), peptic ulcer disease, Gluten Sensitivity and Celiac Disease, Inflammatory Bowel Disease, or history of laparoscopic surgery in GI tract or cholecystectomy.
* Known case of hypertension.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 223 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Stool inflammatory biomarkers | Baseline and 8 weeks
  Change from baseline in myeloperoxidase (MPO)and lipocalin (LCN-2) at 8 weeks measured using ELISA in ng/ml

SECONDARY OUTCOMES:
C-reactive protein (CRP) | Baseline and 8 weeks
  Change from baseline in CRP (mg/ml) at 8 weeks measured using an automated analyzer
Microbiota composition | Baseline and 8 and 12 weeks
  Change from baseline in 16S rRNA (alpha and beta diversity indices) enumeration at 8 and 12 weeks, determined using Illumina-based sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Asad Ali, MPH, Principal Investigator — Aga Khan University Hospital, Karachi
Locations (1):
- Mother and Child Health Research and Training Center, Matiari, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 24 months of study completion
Access Criteria: The Trial Management Group will review data access requests. Requestors will be required to sign a Data Access Agreement.